CLINICAL TRIAL: NCT02345707
Title: A Phase 1, Single-center, Randomized, Open-label, Crossover Study to Assess the Relative Bioavailability of Phase III Tablet Formulation Candidates in Healthy Adult Subjects
Brief Title: Relative Bioavailability Study of Phase III Tablet Formulation of Cabotegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201741
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Cabotegravir; Human Immunodeficiency Virus; Bioavailability; Pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Subjects will receive reference cabotegravir 30 mg current formulation (Treatment A), Cabotegravir 30 mg micronized new formulation 500 M (Treatment B) and Cabotegravir 30 mg unmicronized new formulation 500 U (Treatment C) in one of six sequences ABC, ACB, BCA, BAC, CAB, CBA in three treatment periods under fasting condition
  Interventions: Drug: Cabotegravir 30 mg current formulation; Drug: Cabotegravir 30 mg micronized new formulation 500 M; Drug: Cabotegravir 30 mg unmicronized new formulation 500 U
- Part B (Experimental): Subjects will receive reference Cabotegravir 30 mg current formulation (Treatment A), Cabotegravir 30 mg micronized new formulation 650 M (Treatment D) and Cabotegravir 30 mg unmicronized new formulation 650 U (Treatment E) in one of six sequences ADE, AED, DAE, DEA, EAD, EDA in three treatment periods under fasting condition
  Interventions: Drug: Cabotegravir 30 mg current formulation; Drug: Cabotegravir 30 mg micronized new formulation 650 M; Drug: Cabotegravir 30 mg unmicronized new formulation 650 U

INTERVENTIONS:
Drug: Cabotegravir 30 mg current formulation — Cabotegravir 30 mg current formulation (Treatment A) is a film coated tablet with a weight of 824 mg
Drug: Cabotegravir 30 mg micronized new formulation 500 M — Cabotegravir 30 mg micronized new formulation 500 M (Treatment B) is a film coated tablet with a weight of 515 mg
  Arms: Part A
Drug: Cabotegravir 30 mg unmicronized new formulation 500 U — Cabotegravir 30 mg unmicronized new formulation 500 U (Treatment C) is a film coated tablet with a weight of 515 mg
  Arms: Part A
Drug: Cabotegravir 30 mg micronized new formulation 650 M — Cabotegravir 30 mg micronized new formulation 650 M (Treatment D) is a film coated tablet with a weight of 670 mg
  Arms: Part B
Drug: Cabotegravir 30 mg unmicronized new formulation 650 U — Cabotegravir 30 mg unmicronized new formulation 650 U (Treatment E) is a film coated tablet with a weight of 670 mg
  Arms: Part B

SUMMARY:
This study is a single-center, randomized, open-label, two cohorts, 3-way cross-over design in 36 subjects to assess the oral bioavailability of four new cabotegravir (CAB) sodium salt tablet formulations relative to the current CAB sodium salt formulation being used in the phase IIb studies under fasting conditions. All treatments will be administered as single 30 mg doses of CAB. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 10 - 14 days after the last dose of study drug. Treatment period doses will be separated by a 14 day washout. Participation in this study will be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 18.5 -31.0 kg/ meter square (m^2) (inclusive).
* Male or Female
* Female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies: a) Non-reproductive potential defined as: Pre-menopausal females with one of the following [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy. b) Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause >40 milli-International Units (MIU)/ milliliter (mL) and estradiol <40 picogram (pg)/mL (<147 picomole [pmol]/ liter [L]) is confirmatory]. c) Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until after the last dose of study medication and completion of the follow-up visit. GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP are as follows. This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis. a) Intrauterine device or intrauterine system that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label. b) Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. c) Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository) only for the following 3 situations when there is a very low risk for developmental toxicity: Vaccines; Monoclonal antibodies when there is no target biology concern; Compounds that have a complete reproductive toxicology package and have not shown any signal for developmental toxicity. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. Sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
* Alanine transaminase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of clinically significant cardiovascular disease including: a) Exclusion criteria for screening Electrocardiogram (ECG) (a single repeat is allowed for eligibility determination) Heart rate: Males: <45 and >100 beats per minute, Females: <50 and >100 beats per minute; QRS duration: >120 millisecond (msec), QTc interval (B): >450 msec; b) Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization). c) History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease. d) Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block (AV) block [2nd degree (type II) or higher], Wolf Parkinson White [WPW] syndrome). e) Sinus pauses >3 seconds. f) Any significant arrhythmia which, in the opinion of the principal Investigator and GSK Medical Monitor, will interfere with the safety for the individual subject. g) Non-sustained (>=3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia. NOTES: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial. For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the Reporting and Analysis Plan (RAP).
* Concomitant medications that are prohibited for this study.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Hepatitis B core antibody (HBcAb) with negative hepatitis b surface antibody should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140 millimeters of mercury (mmHg), or diastolic blood pressure is outside the range of 45-90 mmHg.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters for cabotegravir evaluated by measurement of plasma AUC (0-infinity), AUC (0-t) and Cmax and C24 | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120 and 168 hours post dose.
  To evaluate the relative bioavailability of cabotegravir after single 30 mg dose in the fasted state, the following PK parameters will be assessed: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)), area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC (0-t)), maximum observed concentration (Cmax) and concentration at 24 hours post-dose (C24)

SECONDARY OUTCOMES:
Composite of PK parameters for cabotegravir evaluated by measurement of plasma t1/2, tlag, tmax, %AUCex, AUC (0-72), and CL/F | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120 and 168 hours post dose.
  Other plasma PK parameters of cabotegravir from new formulations that will be compared to the current formulation are the following:terminal phase half-life (t ½) , lag time before observation of drug concentrations in sampled matrix (tlag), time of occurrence of Cmax (tmax), percentage of AUC(0-infinity) obtained by extrapolation (%AUCex), area under the concentration-time curve from time zero to 72 hours post dose (AUC (0-72), time of last measurable concentration (tlast) and apparent clearance following oral dosing (CL/F) after single 30 mg dose in the fasted state
Number of participants with adverse events as a measure of safety and tolerability of Cabotegravir | Up to 8 weeks
  Safety and tolerability of cabotegravir will be assessed by clinical safety data from number of participants with adverse event. Adverse events will be collected from the start of study treatment and until the final follow-up visit. Intensity of AEs will be categorized as mild, moderate or severe.
Safety and tolerability of single oral dose of Cabotegravir assessed by concurrent medication used any time during the study period along with the study medication. | Up to 8 weeks
Safety and tolerability of single oral dose of Cabotegravir assessed by clinical laboratory screens | Up to 8 weeks
  Safety laboratory tests will include hematology, clinical chemistry and additional parameters
Safety and tolerability of single oral dose of Cabotegravir assessed by12-lead electrocardiogram | Up to 8 weeks
Safety and tolerability of single oral dose of Cabotegravir assessed by vital signs | Up to 8 weeks
  Vital signs will include systolic and diastolic blood pressure and pulse rate.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States